CLINICAL TRIAL: NCT02827513
Title: A Phase 1 Study to Investigate the Safety, Tolerance, Food Effect, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of Extended Release Formulations of Centanafadine (CTN) (Formerly Called EB-1020) in Young Healthy Subjects
Brief Title: A Phase 1 Study to Investigate the Safety, Tolerance, Food Effect, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of Extended Release Formulations of Centanafadine (CTN) in Young Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVI-EB1020-105
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2016-07

CONDITIONS: Adult Attention-deficit Hyperactivity Disorder (ADHD)
Keywords: Centanafadine; Adult attention-deficit hyperactivity disorder; Healthy participants
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental): Participants will receive sustained release (SR) Tablet Formulation 1 (SR1) containing 100 mg of Centanafadine (CTN) (2 x 100 mg tablets taken orally by mouth [PO] in the morning at starting at approximately 7 am and 2 x 100 mg tablets PO 5 hours later) for a total daily dose (TTD) of 400 mg on Days 1, 4, 7, and 10.
  Interventions: Drug: CTN SR1
- Arm 2 (Experimental): Participants will receive extended release (XR) Tablet Formulation 1 (XR1) containing 400 mg of CTN (1 x 400 mg tablet PO in the morning) on Days 1, 4, 7, and 10.
  Interventions: Drug: CTN XR1
- Arm 3 (Experimental): Participants will receive XR Tablet Formulation 2 (XR2) containing 400 mg of CTN (1 x 400 mg tablet PO in the morning) on Days 1, 4, 7, and 10.
  Interventions: Drug: CTN XR2
- Arm 4 (Experimental): Participants will receive XR Tablet Formulation 3 (XR3) containing 400 mg of CTN (1 x 400 mg tablet PO in the morning) on Days 1, 4, 7, and 10.
  Interventions: Drug: CTN XR3

INTERVENTIONS:
Drug: CTN SR1
  Other Names: Centanafadine
  Arms: Arm 1
Drug: CTN XR1
  Other Names: Centanafadine
  Arms: Arm 2
Drug: CTN XR2
  Other Names: Centanafadine
  Arms: Arm 3
Drug: CTN XR3
  Other Names: Centanafadine
  Arms: Arm 4

SUMMARY:
The purpose of this study is to investigate the safety, tolerance, food effect, pharmacokinetics (PK) and pharmacodynamics (PD) of single and multiple doses of extended release (XR) formulations of Centanafadine (CTN) in Young Healthy participants.

DETAILED DESCRIPTION:
The study will be divided into three parts: A, B, C.

Part A: Single Dose, extended release (XR) Formulation Selection. This part of the study is a single dose, open label, four-period crossover design in a group of 16 healthy participants.

Part B: Multiple Ascending Dose. Part B has been designed to assess the effect of multiple doses of one formulation of XR CTN. This part of the study will be a double-blind, randomized, placebo-controlled design.

Part C: Food Effect. Part C has been designed to determine the effect food has on XR CTN. The XR formulation and dose administered will be selected after review of Part B data. This part will be an open-label, two-period crossover design in a group of 16 healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Body weight within the normal range for height (body mass index [BMI] between 19-30 kg/m2 inclusive);
2. Negative serum pregnancy test at Screening and negative urine pregnancy test at Day -1 for females of child bearing potential;
3. Women of child-bearing potential must agree to use adequate; contraception prior to study entry, for the duration of study participation, and for 90 days following completion of therapy;
4. Be in general good health without clinically significant medical history;
5. Have clinical laboratory test results that are within the laboratory reference range; or if out of range are not clinically relevant and are acceptable to the Investigator and Sponsor medical representative;
6. Negative Human Immunodeficiency Virus (HIV), Hepatitis B and Hepatitis C Screening test;
7. Able and willing to give written informed consent.

Exclusion Criteria:

1. Use of any of the following medications will exclude a participant:

   * investigational compound within 30 days prior to Screening;
   * antipsychotic, anxiolytic, or sedative-hypnotic medication within 30 days prior to Screening;
   * any antidepressant medication within 30 days prior to Screening;
   * clonidine within 30 days prior to Screening;
   * cough/cold preparations containing stimulants/sympathomimetic agent within 7 days prior to Day -1;
   * norepinephrine reuptake inhibitors, such as tomoxetine (STRATTERA®) within 30 days prior to Day -1;
   * antihypertensive agents, including diuretics, are not permitted at any time prior to or during the study;
   * sedating antihistamines (as a single preparation or in combination) within 7 days prior to Day -1;
   * sympathomimetics, appetite suppressants, modafinil, methylphenidate, amphetamine and pemoline within 7 days prior to Day -1;
   * Use over the counter medications within 7 days of Investigational Product administration, with the exception of simple analgesics such as paracetamol, oral non-steroidal anti-inflammatory agents and the oral contraceptive pill (if applicable);
   * Use of any herbal preparations and melatonin is prohibited and should be discontinued prior to Day -1. The process for discontinuing use of herbal preparations and melatonin prior to Day -1 is at the discretion of the Investigator;
2. A history of, or current evidence for, suicidal ideation, based upon clinical interview and the Columbia Suicide Severity Rating Scale (C-SSRS);
3. A history of known or suspected seizures, spasms, infantile spasms, febrile convulsions, unexplained significant and recent loss of consciousness or history of significant head trauma with loss of consciousness or a family history (first degree relative) of epilepsy or seizures (fits);
4. Subject has a known history of hypertension or Subject has a supine systolic blood pressure (SBP) ≥140 mm Hg or diastolic blood pressure (DBP) ≥90 mm Hg. No more than one repeat measurement will be permitted;
5. Subject has a known history of orthostatic hypotension or has an orthostatic blood pressure (BP) drop of ≥20 mm Hg (based on the drop between supine and standing [3 minutes] SBP) at Screening or Day -1;

Note: The eligibility criteria list is not exhaustive.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events and serious adverse events | Up to approximately 12 days

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of Centanafadine (CTN) and metabolite | For Part A: From Day 1 to 12; For Part B: Day 1, Day 2, Day 4, Day 5, Day 6, and Day 7; For Part C: Day 1 to 6
  Blood samples for the determination of plasma concentrations of CTN and metabolite will be collected following dosing as follows: For Part A- on Days 1, 4, 7, and 10 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 18; Days 2, 5, 8, and 11 at hour 24, 30, and 36; Days 3, 6, 9, and 12 at hour 48. For Part B- on Day 1 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 2 at Hour 24/Pre-dose; Day 4 at Pre-dose; Day 5 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 6 at hour 24 and 36; Day 7 at hour 48. For Part C- on Days 1 and 4 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 18; Days 2 and 5 at hour 24, 30, and 36; Days 3 and 6 at hour 48
Time to maximum plasma concentration (Tmax) of CTN and metabolite | For Part A: From Day 1 to 12; For Part B: Day 1, Day 2, Day 4, Day 5, Day 6, and Day 7; For Part C: Day 1 to 6
  Blood samples for the determination of plasma concentrations of CTN and metabolite will be collected following dosing as follows: For Part A- on Days 1, 4, 7, and 10 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 18; Days 2, 5, 8, and 11 at hour 24, 30, and 36; Days 3, 6, 9, and 12 at hour 48. For Part B- on Day 1 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 2 at Hour 24/Pre-dose; Day 4 at Pre-dose; Day 5 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 6 at hour 24 and 36; Day 7 at hour 48. For Part C- on Days 1 and 4 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 18; Days 2 and 5 at hour 24, 30, and 36; Days 3 and 6 at hour 48
Area under the plasma concentration-time curve from time zero until the last quantifiable time point (AUC0-last) of CTN and metabolite | For Part A: From Day 1 to 12; For Part B: Day 1, Day 2, Day 4, Day 5, Day 6, and Day 7; For Part C: Day 1 to 6
  Blood samples for the determination of plasma concentrations of CTN and metabolite will be collected following dosing as follows: For Part A- on Days 1, 4, 7, and 10 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 18; Days 2, 5, 8, and 11 at hour 24, 30, and 36; Days 3, 6, 9, and 12 at hour 48. For Part B- on Day 1 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 2 at Hour 24/Pre-dose; Day 4 at Pre-dose; Day 5 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 6 at hour 24 and 36; Day 7 at hour 48. For Part C- on Days 1 and 4 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 18; Days 2 and 5 at hour 24, 30, and 36; Days 3 and 6 at hour 48
Apparent termination elimination rate constant (kel) of CTN and metabolite | For Part A: From Day 1 to 12; For Part B: Day 1, Day 2, Day 4, Day 5, Day 6, and Day 7; For Part C: Day 1 to 6
  Blood samples for the determination of plasma concentrations of CTN and metabolite will be collected following dosing as follows: For Part A- on Days 1, 4, 7, and 10 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 18; Days 2, 5, 8, and 11 at hour 24, 30, and 36; Days 3, 6, 9, and 12 at hour 48. For Part B- on Day 1 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 2 at Hour 24/Pre-dose; Day 4 at Pre-dose; Day 5 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 6 at hour 24 and 36; Day 7 at hour 48. For Part C- on Days 1 and 4 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 18; Days 2 and 5 at hour 24, 30, and 36; Days 3 and 6 at hour 48
Apparent terminal elimination half-life (t1/2) of CTN and metabolite | For Part A: From Day 1 to 12; For Part B: Day 1, Day 2, Day 4, Day 5, Day 6, and Day 7; For Part C: Day 1 to 6
  Blood samples for the determination of plasma concentrations of CTN and metabolite will be collected following dosing as follows: For Part A- on Days 1, 4, 7, and 10 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 18; Days 2, 5, 8, and 11 at hour 24, 30, and 36; Days 3, 6, 9, and 12 at hour 48. For Part B- on Day 1 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 2 at Hour 24/Pre-dose; Day 4 at Pre-dose; Day 5 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 6 at hour 24 and 36; Day 7 at hour 48. For Part C- on Days 1 and 4 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 18; Days 2 and 5 at hour 24, 30, and 36; Days 3 and 6 at hour 48
last measurable plasma concentration (Clast) of CTN and metabolite | For Part A: From Day 1 to 12; For Part B: Day 1, Day 2, Day 4, Day 5, Day 6, and Day 7; For Part C: Day 1 to 6
  Blood samples for the determination of plasma concentrations of CTN and metabolite will be collected following dosing as follows: For Part A- on Days 1, 4, 7, and 10 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 18; Days 2, 5, 8, and 11 at hour 24, 30, and 36; Days 3, 6, 9, and 12 at hour 48. For Part B- on Day 1 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 2 at Hour 24/Pre-dose; Day 4 at Pre-dose; Day 5 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 6 at hour 24 and 36; Day 7 at hour 48. For Part C- on Days 1 and 4 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 18; Days 2 and 5 at hour 24, 30, and 36; Days 3 and 6 at hour 48
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) from AUC0-last +Clast/kel of CTN and metabolite | For Part A: From Day 1 to 12; For Part B: Day 1, Day 2, Day 4, Day 5, Day 6, and Day 7; For Part C: Day 1 to 6
  Blood samples for the determination of plasma concentrations of CTN and metabolite will be collected following dosing as follows: For Part A- on Days 1, 4, 7, and 10 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 18; Days 2, 5, 8, and 11 at hour 24, 30, and 36; Days 3, 6, 9, and 12 at hour 48. For Part B- on Day 1 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 2 at Hour 24/Pre-dose; Day 4 at Pre-dose; Day 5 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 6 at hour 24 and 36; Day 7 at hour 48. For Part C- on Days 1 and 4 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 18; Days 2 and 5 at hour 24, 30, and 36; Days 3 and 6 at hour 48
Dose normalized Cmax (Cmax/Dose) of CTN and metabolite | For Part A: From Day 1 to 12; For Part B: Day 1, Day 2, Day 4, Day 5, Day 6, and Day 7; For Part C: Day 1 to 6
  Blood samples for the determination of plasma concentrations of CTN and metabolite will be collected following dosing as follows: For Part A- on Days 1, 4, 7, and 10 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 18; Days 2, 5, 8, and 11 at hour 24, 30, and 36; Days 3, 6, 9, and 12 at hour 48. For Part B- on Day 1 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 2 at Hour 24/Pre-dose; Day 4 at Pre-dose; Day 5 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 6 at hour 24 and 36; Day 7 at hour 48. For Part C- on Days 1 and 4 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 18; Days 2 and 5 at hour 24, 30, and 36; Days 3 and 6 at hour 48
Dose normalized AUC (AUC/Dose) of CTN and metabolite | For Part A: From Day 1 to 12; For Part B: Day 1, Day 2, Day 4, Day 5, Day 6, and Day 7; For Part C: Day 1 to 6
  Blood samples for the determination of plasma concentrations of CTN and metabolite will be collected following dosing as follows: For Part A- on Days 1, 4, 7, and 10 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 18; Days 2, 5, 8, and 11 at hour 24, 30, and 36; Days 3, 6, 9, and 12 at hour 48. For Part B- on Day 1 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 2 at Hour 24/Pre-dose; Day 4 at Pre-dose; Day 5 at Pre-dose, hour 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 18; Day 6 at hour 24 and 36; Day 7 at hour 48. For Part C- on Days 1 and 4 at Pre-dose, hour 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 18; Days 2 and 5 at hour 24, 30, and 36; Days 3 and 6 at hour 48

CONTACTS AND LOCATIONS:
Locations (1):
- Melbourne, Australia